CLINICAL TRIAL: NCT04203355
Title: Multi-country, Multi-center Cohort Study of Anti-Mullerian Hormone Profile in Asia Pacific Infertile Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: TMU201912130
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to detect the infertile couple (women) Anti-Mullerian Hormone (AMH) profile in major subgroups such as Poly Cystic Ovarian Syndrome (PCOS), Endometriosis, etc via age intervals and ethnic difference.

DETAILED DESCRIPTION:
To consecutively enroll infertile couple (women) who are undergoing their first controlled ovarian stimulation cycles.

To mainly compare the inter-ethnic difference in age-specific AMH profile in unexplained infertility, male factor infertility, PCOS, Endometriosis etc. subgroups.

To detect the influence of past or present smoking on age-specific AMH levels To study the influence of body mass index (BMI) on age specific AMH levels

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as infertile couple
* Naive patients who plan to enter their first ovarian stimulation cycles
* Women among 20-43 years old

Exclusion Criteria:

* Systematic disease that impact AMH (eg. systemic lupus erythematosus (SLE), Crohn's disease etc.)
* Chemotherapy history
* Alcohol abuse
* Currently taking oral contraceptive pills

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Those diagnosed as infertile couples (male or female infertility) and plan to enter their first ovarian stimulation cycles. Those women are 20-43 years old are enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Anti-mullerian hormone level in general population | within 3 months before controlled ovarian stimulation cycles
  Inter-ethnic difference in age-specific AMH level

SECONDARY OUTCOMES:
Anti-mullerian hormone level in PCOS patients | within 3 months before controlled ovarian stimulation cycles
  AMH level in PCOS patients vs non-PCOS patients in age-specific intervals
Anti-mullerian hormone level in endometriosis patients | within 3 months before controlled ovarian stimulation cycles
  AMH level in endometriosis patients vs non-endometriosis patients in age-specific intervals

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Ruey Tzeng, MD, Ph.D, Principal Investigator — Taipei Medical University Hospital
Locations (11):
- Henan Provincial People Hospital, Zhengzhou, Henan, China
- Queen Mary Hospital, Hong Kong, Hong Kong
- Women's center by Motherhood Coimbatore, Bangalore, Karnataka, India
- Morula IVF center, Jakarta, Indonesia
- Asada Ladies Clinic, Nagoya, Aichi-ken, Japan
- Tropicana Medical Centre, Petaling Jaya, Selangor, Malaysia
- Victory ART Lab Fertility Center, Makati City, Philippines
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea
- Taipei University Medical Hospital, Taipei, Taiwan
- Chiang Mai University, Chiang Mai, Thailand
- My Duc Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Tzeng CR, Huang Z, Asada Y, Zhang C, Ho MT, Li RHW, Kim JH, Govindarajan M, Vuyavanich T, Sini I, Wong PS, Singh S, Lin WY, Ho NT. Factors affecting the distribution of serum anti-mullerian hormone levels among infertile Asian women: a multi-nation, multi-centre, and multi-ethnicity prospective cohort study. Hum Reprod. 2023 Jul 5;38(7):1368-1378. doi: 10.1093/humrep/dead081. PMID 37105234